CLINICAL TRIAL: NCT05855070
Title: Intralesional Injection of Hyaluronic Acid Compared With Verapamil in Peyronie's Disease: A Prospective Randomized Clinical Trial
Brief Title: Intralesional Hyaluronic Acid and Verapamil Injection in Peyronie's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abou Elezz Abdel Fattah, Lecturer of Urology, Faculty of Medicine, Benha University, Benha, Egypt, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC 6-5-2023
Record Dates: First submitted 2023-05-03; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Peyronie's Disease; Hyaluronic Acid; Verapamil
MeSH Terms: conditions — Penile Induration | interventions — Hyaluronic Acid; Verapamil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intralesional treatment with Hyaluronic acid (Experimental): Patients will receive intralesional treatment with Hyaluronic acid (0.8% highly purified sodium salt Hyaluronic acid 6 mg/2 mL; Sinovial, IBSA, Lodi, Italy) weekly for 12 weeks.
  Interventions: Drug: Intralesional treatment with Hyaluronic acid
- Intralesional treatment with Verapamil (Experimental): Patients will receive intralesional treatment with Verapamil (10 mg in 5 mL of normal saline water) weekly for 12 weeks.
  Interventions: Drug: Intralesional treatment with Verapamil

INTERVENTIONS:
Drug: Intralesional treatment with Hyaluronic acid — Patients will receive intralesional treatment with Hyaluronic acid (0.8% highly purified sodium salt Hyaluronic acid16 mg/2 mL; Sinovial, IBSA, Lodi, Italy) weekly for 12 weeks.
  Arms: Intralesional treatment with Hyaluronic acid
Drug: Intralesional treatment with Verapamil — Patients will receive intralesional treatment with Verapamil (10 mg in 5 mL of normal saline water) weekly for 12 weeks.
  Arms: Intralesional treatment with Verapamil

SUMMARY:
The aim of the present study is to investigate whether intralesional injections of Hyaluronic acid in the acute phase could reduce the progression of Peyronie's disease thanks to its interference with inflammatory and pro-fibrotic processes.

Therefore, a prospective, longitudinal, double-blinded, randomized clinical study, has been designed to evaluate and compare the efficacy and safety of intralesional HA as compared with the use of verapamil injection in patients affected by Peyronie's disease.

DETAILED DESCRIPTION:
Peyronie's disease is defined as a chronic benign condition characterized by the formation of localized fibrous inelastic scars at the level of the tunica albuginea of the penis. This condition can lead to penile curvature, painful erections and erectile dysfunction. Peyronie's disease is believed to affect 3% to 9% of the male population, with a higher prevalence among patients suffering from erectile dysfunction, diabetes and cardiovascular disease .

The etiology of Peyronie's disease is largely unknown. According to current popular theories, a single traumatic event or repeated microtraumas during sexual activity can lead to a low-level autoimmune response arising from a prolonged and complex inflammatory reaction of the tunica albuginea fibers,5 which leads to plaque formation.

The Peyronie's disease presents 2 different phases: active or acute and stable or chronic. It is paramount to distinguish between acute and chronic phase of the condition, since management is different in the 2 phases. Plaque formation and calcification generally take place during the acute phase, which can last for up to 18 months. In the chronic phase, penile pain will be reduced, and penile deformity stabilized. Transition to the chronic phase is defined when curvature remains stable for at least 3 months.

The European Association of Urology and the American Association of Urology have released clinical practice guidelines for the diagnosis, evaluation, treatment, and follow-up of patients with Peyronie's disease.

Treatment of Peyronie's disease includes both medical and surgical approaches and the management is tailored to the phase of the disease, the degree of deformity, the quality of the erections and patient's choice.

Conservative treatment of Peyronie's disease is focused primarily on patients in the early (acute inflammatory) stage, and surgical remediation is used to correct curvature, allow for satisfactory intercourse, and is reserved for patients who have stable disease for at least 12 months .

ELIGIBILITY:
Inclusion Criteria:

* Patient's age from >18 - 70 years old.
* A palpable nodule or plaque in the tunica of the penis
* Presence of pain in the flaccid state or during painful erections.
* Progressive penile curvature >15° and/or penile pain in the flaccid state or at the erection in the last 12 months

Exclusion Criteria:

* Patient refusal.
* Calcified plaques or hourglass deformity as defined at duplex Doppler ultrasonography,
* Previous Peyronie's Disease therapy with oral agents or intralesional injections
* Severe concomitant erectile dysfunction (International Index of Erectile Function [IIEF-5] score < 7).
* Congenital penile curvature, history of previous penile surgery, a concomitant oral treatment for Peyronie's Disease.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Sexually active men older than 18 years affected by Peyronie's Disease
Enrollment: 42 (Estimated)
Dates: Start 2023-05-20 (Estimated); Primary Completion 2024-05-20 (Estimated); Study Completion 2024-05-20 (Estimated)

PRIMARY OUTCOMES:
Penile curvature degree | 12 weeks postoperatively
  The change from the baseline to the endpoint (12 weeks after therapy) for the penile curvature (degree).

SECONDARY OUTCOMES:
Plaque size (mm) | 12 weeks postoperatively
  The change in plaque size (mm) will be recorded

IPD SHARING:
Plan to Share IPD: Yes
The study will be available under a reasonable request from the corresponding author.
Supporting Information: Study Protocol
Time Frame: One year after the end of the study.